CLINICAL TRIAL: NCT02525315
Title: Interest of Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of Auditory Hallucinations
Acronym: TMS HALLU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-137
Record Dates: First submitted 2015-08-13; First posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Schizophrenic Disorders
Keywords: Schizophrenia; auditory hallucinations; TMS
MeSH Terms: conditions — Schizophrenia; Hallucinations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transcranial magnetic stimulation: rTMS (Experimental): rTMS : 4 sessions of 13 minutes, with 2 sessions a day, at 20Hz frequency and at an intensity of 80% of rest motor threshold will be delivered
  Interventions: Device: Transcranial magnetic stimulation: rTMS

INTERVENTIONS:
Device: Transcranial magnetic stimulation: rTMS — 4 sessions of 13 minutes, with 2 sessions a day, at 20Hz frequency and at an intensity of 80% of rest motor threshold will be delivered

SUMMARY:
Auditory hallucinations are common (present in 60-70% of cases) and extremely debilitating. Behavioral disorders associated with them can have serious social repercussions. However, in 25% of cases the usual antipsychotic drug treatments are incompletely or totally ineffective.

Fifteen subjects will be included after collection and signed their informed consent.

The rTMS treatment is made of 4 sessions of 13 minutes spread over two days, at a frequency of 20 Hz and an intensity of 80% of motor threshold at rest. These constants are used to stay below the risk of occurrence of seizures, the only serious side effects identified. Furthermore the rTMS treatment is almost painless: tension headaches are the main side effects and make amends with simple analgesics. rTMS is devoid of neurocognitive effects. The LEFT stimulation site will be established through a anatomofunctional imaging before treatment (between D-7 and D0).

Treatment efficacy will be evaluated daily during treatment (days 1 and 2) and during the first 2 weeks of starting treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenic disorders aged from 18 to 60 years old
* Patients suffering from auditory hallucinations undergoing antipsychotic treatments
* Written signed consent

Exclusion Criteria:

* Pregnancy or breastfeeding
* Counter-indication to MRI or to rTMS

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2007-06; Primary Completion 2012-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
HOFFMAN score | change between baseline and day 3 or day 12

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Dollfus, MD, PhD, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, France